CLINICAL TRIAL: NCT04462211
Title: Pilot Study of the Preparation and Implementation of a Constipation Bundle & Management Protocol and the Effect of Adherence in Reducing the Incidence of Constipation in Critically Ill Patients of a University Hospital
Brief Title: Constipation Bundle/Protocol and the Effect of Adherence in the Incidence of Constipation in Critically Ill Patients
Acronym: motility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Tobar, Associated Professor, University of Chile
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OAIC1055/19
Record Dates: First submitted 2019-12-19; First posted 2020-07-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Constipation; Critical Illness; Constipation Drug Induced
MeSH Terms: conditions — Constipation; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Management pharmacological protocol and bundle's (Experimental): The elaboration of the protocol according to the evidence-based approach, updated evidence found from both search engines such as MEDLINE, EMBASE, Cochrane Library, OVID and ScIELO will be used through the research question using the PICO method (Patient interest, Intervention, Comparation and Outcome).
  the ready-made protocol will be adjusted to the pharmacological options that are available in the hospital.
  Interventions: Procedure: Implementation of management pharmacological protocol of constipation; Procedure: Implementation of bundle of prevention and non-pharmacological management

INTERVENTIONS:
Procedure: Implementation of management pharmacological protocol of constipation — first 48 hours:
  * polyethylene glycol 3350 (about 17 grams) 1 every 8 hours enterally.
  * Patients who have vomiting and / or gastric residue greater than 500 mL (in a timely measurement every 6 hours) will also be given domperidone 10 mg every 8 hours intravenously.
  * Patients who have excessive abdominal distension will be administered in addition, levosulpiride 25 mg every 8 hours intravenously.
    48 hour evaluation:
  * Patients who do not have bowel movements will be administered lactulose or sodium phosphate enema.
  * For patients who do not have a bowel movement, administration of neostigmine intravenously or of naloxone enterally will be evaluated.
  * Every patient who uses one or more prokinetics will have an electrocardiogram.
  * Any patient who has bowel movements during management, doses of polyethylene glycol 3350 will be adjusted according to the daily goal of bowel movements, the days of treatment of the prokinetics will be adjusted, for a maximum of 5 consecutive days.
Procedure: Implementation of bundle of prevention and non-pharmacological management — Bundle of prevention:
  * Start early enteral nutrition.
  * Optimize and / or decrease opioid doses.
  * Start early mobilization.
  Non-pharmacological management bundle
  * Select laxative and/or prokinetic/s to manage constipation.
  * Optimize and / or decrease doses of opioids and sedatives.
  * Start early mobilization.
  * Pharmacological reconciliation.

SUMMARY:
Gastrointestinal abnormalities are present in more than 80% of critical patients, and their management has taken an important importance in intensive care unit (ICU), since it can largely determine the clinical outcome, costs and long-term prognosis in This group of patients. Only the constipation in the critical patient has been related to the failure of weaning of the mechanical ventilator, an increase in mechanical ventilation time, and with the increase of the stay in the ICU.

In general, most critical health conditions cause a decrease in the motility of the gastrointestinal tract that intrinsically can contribute to constipation. This is explained by the increase in pro-inflammatory cytokines, increased activity of the sympathetic system, the use of vasopressors, high and prolonged doses of opiates, among others, which can reduce gastric emptying and delay motility. These gastrointestinal abnormalities may be associated with an increase in intra-abdominal pressure, reduced nutritional intake, bacterial hyperproliferation in the digestive tract, intestinal mucosal injury and bacterial translocation through the injured and / or inflamed mucosa. In addition, patients who experience constipation often have gastroparesis and paresis of the ileum, conditions that hinder the progression of nutritional support enterally and worsen the patient's clinical picture.

In spite of being quite common in the ICU, the impact is not known in depth, which implies that these alterations are usually not prevented and on the other hand when treating their pharmacological and non-pharmacological management is highly variable because, for a On the other hand, staff turnover (intensivist physician) and on the other hand because there are no protocols that reduce these problems.

To provide comprehensive care in critical patient units, according to the best available evidence in order to reduce the variation in daily care, clinical guidelines and protocols are applied to manage the various specific problems that affect this group. of patients One way to address the complexity of these problems is through the implementation of care packages, which have taken relevance in the prevention of characteristic events of high mortality and morbidity. It is in this scenario, where the clinical pharmacist plays an important role in the development of protocols, packages and their compliance. The clinical pharmacist is dedicated to the review of the therapy of each patient, through pharmacological conciliation actions with the attending physician, actively participating in the daily round of the multidisciplinary team and at the same time developing "professional support activities" that include , reviews of adverse events associated with medications, education, auditing, research, development of guidelines and institutional protocols for the use of effective and safe medications, with the objective of reducing mortality and its associated costs, thus improving the quality of the Attention.

Given the importance of the problem, it is that this work proposes that the implementation and active dissemination of a constipation bundle/protocol guided by a clinical pharmacist ensures adherence to the strategy in the treatment team and a decrease in the incidence of constipation in the critical patient of the ICU of a university hospital. To fulfill this objective, a quasi-experimental study was designed in which the first stage will be diagnostic observational and a second part of the interventional type, in order to evaluate the effect of adherence to the bundle/protocol on the incidence of constipation in critically ill patients admitted to a ICU of a university hospital for a period of 6 months.

DETAILED DESCRIPTION:
Stages of the study

The project will be carried out in 5 phases distributed in 3 continuous periods of time.

* Stage 1 - 2 month period (observational period).
* Collection of patient information for bundle/protocol development.
* Stage 2 - 3 month period.
* Protocol / bundle development according to evidence-based approach
* Active dissemination of bundle/protocol.
* Stage 3 - 1 month period (implementation and evaluation period)
* Protocol / bundle implementation.
* Collection of patient information, measurement of adherence and evaluation of the effect of the bundle/protocol.

Description of the Phases of the Study

Stage 1

• Collection of patient information for the elaboration of the bundle/protocol.

Information from patients hospitalized at the ICU will be collected through a data collection sheet, prospectively to quantify the local magnitude of the constipation and other alterations associated with the decrease in intestinal motility, interventions performed with their results and its consequences.

The data will be collected through a collection form, which will consist of 5 parts:

* Part I: Basic background record (Age, gender, anthropometric data, ICU service you enter, service from which it comes, chronic morbid history).
* Part II: Registration of factors in the patient that may be related to the presence of gastrointestinal motility disorders, as a risk or protective factor during the stay in ICU (type of mechanical ventilation, use of norepinephrine, medicines used in sedoanalgesia, degree of sedation according to SAS scale)
* Part III: Characterization of the nutrition administered to the patient during the stay in ICU (what type of enteral nutrition he is receiving, daily amount of nutrition, daily water balance, amount of bowel movements and if he has diarrhea).
* Part IV: Registry of Laxative/s and/or Prokinetic/s Treatment and its clinical evolution.
* Part V: Identification and Registration of adverse effects associated with the indicated treatment that are clinically evaluable and/or by registration in the nursing and medical record.

Stage 2

• Bundle/protocol development according to evidence-based approach

Protocol and bundle elaboration.

• Active dissemination of a constipation protocol / bundle.

Implementation strategies will be addressed using the EPOC taxonomy (Effective Practice and Organization of Care (EPOC). EPOC taxonomy. Oslo: Norwegian Knowledge Center for the Health Services; 2002). For the purpose of this work only part of the

Interventions aimed at health professionals.

A. Distribution of the protocol and bundles by email and a hard copy to all unit heads. In addition, all the professional prescribers of the unit will be given a hard copy.

B. Educational Talks: Directed to health professionals.

* Active education: Session in groups of no more than 10 people, usually carried out in medical visits, as feedback in multidisciplinary reviews of a patient between different professionals of the medical team and/or interconsultores (professionals from other disciplines and/or units other than within the ICU), in order to engage and educate the health professional about the interventions of the protoco and the bundles, and also confirm learning by the professional.
* Passive education: Sessions intended to disseminate information to the prescribing doctors of the entire unit, and to solve doubts globally.

C. Local opinion leaders:

Intervention through the participation of health professionals designated by their colleagues as "educationally influential" (health professionals staff of the ICU, nutritionist, gastroenterologist or others)

D. Reminders: any oral or visual intervention that encourages the health professional to perform a clinical action related to the protocol / bundle. The following interventions are included:

* Oral reminders (Aimed at both treating physician, medical staff, and nurse between medical visits when there is evidence of suboptimal care for patients included in the study, for example, when a patient is constipated and is not receiving treatment).
* Administrative support (graphics or reminder stickers attached to each patient's box).

Organizational Interventions:

A. Structural interventions Incorporation of the protocol and bundles in each medical record of the patients included.

Stage 3

• Implementation of the bundle/protocol in patients admitted during this period, who meet the inclusion criteria and our treating doctors accepted informed consent (if necessary).

The patients included in phase 3 of the study corresponding to the implementation of the package will be patients of the ICU, whatever the applications during the statistics, the set of exclusive controls for each service unit (previously accepted as a package) focused on the prevention of a probable episode of constipation, as long as there is no contraindication (previously described). If a patient included in the corresponding phase of the study will present constipation, the pharmacological management for said health problem will be applied, as specified in their "pharmacological management protocol for constipation" developed and validated together with the package.

These protocol / package interventions will be presented to the health team during medical rounds by both the pharmaceutical chemist responsible for the investigation and by any other professional of the patient's health team in order to comply with the adherence to the protocol / package for each patient

• Collection of patient information, adherence measurement and evaluation of the effect of the protocol / package.

Information from hospitalized patients in the ICU will be collected through a data collection form previously validated in Stage 1. In addition, the following information will be incorporated:

* Part I to Part V: Identical to the one previously validated.
* Part VI: Applicability of bundle in each of the elements.
* Part VII: Applicability of protocol.

This data will be backed up in an EXCEL (office) format file for later analysis.

Sample size

The universe and the target population will be all admitted patients that meet the inclusion criteria in the period of time in which stage 1 (observational period) and stage 3 (period of implementation and evaluation) of the study are executed

Events to evaluate

In this research paper:

The effectiveness of the analysis of the following definitions shall be understood:

• Adhesion: It will be understood as adherence to the effective fulfillment of the interventions that will be prepared for the protocol and the bundle.

• Constipation: Constipation shall be understood as the presence of "three or more consecutive days without depositions" and prolonged constipation as "six or more consecutive days without depositions". For both definitions, it will be considered as zero day without depositions from the start of enteral nutrition, at most 96 hours after admission to the ICU.

Safety shall be understood as the analysis of adverse events described in the following definitions:

• Intolerance to nutritional support: It is understood as an intolerance to enteral nutritional support to the presence of "gastric residue greater than 500mL in a measurement during the day, or to the presence of vomiting", which will be taken into account in patients who are being given enteral nutrition.

• Liquid deposition: Liquid deposition shall be understood as the presence of a "deposition of liquid consistency quantified in an amount greater than 200 milliliters". It is also synonymous with a diarrheal deposition. *

• Mechanical fan day: A mechanical ventilator day will be considered when the patient requires mechanical ventilator support for more than 12 hours on the day of hospitalization analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the intensivo care unit.
* Hospitalization equal to or greater than 3 days.

Exclusion Criteria:

* Patient admitted after surgery for resection of the digestive tract.
* Patient with exclusive parenteral nutrition.
* Patient with total intestinal obstruction / ileus, documented during the stay at UPC.
* Patients admitted exclusively for "isolation measures".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Adherence to protocol / bundle implementation. | 1 mounth
  The adherence for the protocol and for the bundle will be evaluated by being separated. Both will be evaluated by dichotomous evaluation (is adherent or not adherent). It is adherent for the bundle only if all the interventions for the bundle are fulfilled, likewise, it is adherent for the protocol if all the interventions for the protocol are fulfilled.

SECONDARY OUTCOMES:
Difference in incidence of constipation between observational period group and protocol / bundle implementation period group. | 1 mounths.
  Constipation is assessed using the described definition, every day.
Intolerance to nutritional. | 1 mounths
  All presence of "gastric residue greater than 500mL in a measurement during the day, or to the presence of vomiting" will be recorded.
Liquid deposition. | 1 mounths.
  all presence of a "deposition of liquid consistency quantified in an amount greater than 200 milliliters" will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: José Ignacio JI Farías, Pharmacist, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, International, Chile

REFERENCES:
- [Background] Reintam Blaser A, Malbrain ML, Starkopf J, Fruhwald S, Jakob SM, De Waele J, Braun JP, Poeze M, Spies C. Gastrointestinal function in intensive care patients: terminology, definitions and management. Recommendations of the ESICM Working Group on Abdominal Problems. Intensive Care Med. 2012 Mar;38(3):384-94. doi: 10.1007/s00134-011-2459-y. Epub 2012 Feb 7. PMID 22310869
- [Background] Rohm KD, Boldt J, Piper SN. Motility disorders in the ICU: recent therapeutic options and clinical practice. Curr Opin Clin Nutr Metab Care. 2009 Mar;12(2):161-7. doi: 10.1097/MCO.0b013e32832182c4. PMID 19202387
- [Background] Btaiche IF, Chan LN, Pleva M, Kraft MD. Critical illness, gastrointestinal complications, and medication therapy during enteral feeding in critically ill adult patients. Nutr Clin Pract. 2010 Feb;25(1):32-49. doi: 10.1177/0884533609357565. PMID 20130156
- [Background] Gacouin A, Camus C, Gros A, Isslame S, Marque S, Lavoue S, Chimot L, Donnio PY, Le Tulzo Y. Constipation in long-term ventilated patients: associated factors and impact on intensive care unit outcomes. Crit Care Med. 2010 Oct;38(10):1933-8. doi: 10.1097/CCM.0b013e3181eb9236. PMID 20639749
- [Background] Prat D, Messika J, Millereux M, Gouezel C, Hamzaoui O, Demars N, Jacobs F, Trouiller P, Ricard JD, Sztrymf B. Constipation in critical care patients: both timing and duration matter. Eur J Gastroenterol Hepatol. 2018 Sep;30(9):1003-1008. doi: 10.1097/MEG.0000000000001165. PMID 29794547
- [Background] Prat D, Messika J, Avenel A, Jacobs F, Fichet J, Lemeur M, Ricard JD, Sztrymf B. Constipation incidence and impact in medical critical care patients: importance of the definition criterion. Eur J Gastroenterol Hepatol. 2016 Mar;28(3):290-6. doi: 10.1097/MEG.0000000000000543. PMID 26709885
- [Background] Taylor RW. Gut Motility Issues in Critical Illness. Crit Care Clin. 2016 Apr;32(2):191-201. doi: 10.1016/j.ccc.2015.11.003. Epub 2016 Feb 18. PMID 27016161
- [Background] Ukleja A. Altered GI motility in critically Ill patients: current understanding of pathophysiology, clinical impact, and diagnostic approach. Nutr Clin Pract. 2010 Feb;25(1):16-25. doi: 10.1177/0884533609357568. PMID 20130154
- [Background] Fruhwald S, Holzer P, Metzler H. Intestinal motility disturbances in intensive care patients pathogenesis and clinical impact. Intensive Care Med. 2007 Jan;33(1):36-44. doi: 10.1007/s00134-006-0452-7. Epub 2006 Nov 18. PMID 17115132
- [Background] Mostafa SM, Bhandari S, Ritchie G, Gratton N, Wenstone R. Constipation and its implications in the critically ill patient. Br J Anaesth. 2003 Dec;91(6):815-9. doi: 10.1093/bja/aeg275. PMID 14633751
- [Background] Nassar AP Jr, da Silva FM, de Cleva R. Constipation in intensive care unit: incidence and risk factors. J Crit Care. 2009 Dec;24(4):630.e9-12. doi: 10.1016/j.jcrc.2009.03.007. Epub 2009 Jul 9. PMID 19592200
- [Background] Patanwala AE, Abarca J, Huckleberry Y, Erstad BL. Pharmacologic management of constipation in the critically ill patient. Pharmacotherapy. 2006 Jul;26(7):896-902. doi: 10.1592/phco.26.7.896. PMID 16803421
- [Background] de Azevedo RP, Machado FR. Constipation in critically ill patients: much more than we imagine. Rev Bras Ter Intensiva. 2013 Apr-Jun;25(2):73-4. doi: 10.5935/0103-507X.20130014. No abstract available. PMID 23917968
- [Background] Farmer AD, Holt CB, Downes TJ, Ruggeri E, Del Vecchio S, De Giorgio R. Pathophysiology, diagnosis, and management of opioid-induced constipation. Lancet Gastroenterol Hepatol. 2018 Mar;3(3):203-212. doi: 10.1016/S2468-1253(18)30008-6. PMID 29870734
- [Background] McPeake J, Gilmour H, MacIntosh G. The implementation of a bowel management protocol in an adult intensive care unit. Nurs Crit Care. 2011 Sep-Oct;16(5):235-42. doi: 10.1111/j.1478-5153.2011.00451.x. PMID 21824228
- [Background] Borgert M, Binnekade J, Paulus F, Goossens A, Dongelmans D. A flowchart for building evidence-based care bundles in intensive care: based on a systematic review. Int J Qual Health Care. 2017 Apr 1;29(2):163-175. doi: 10.1093/intqhc/mzx009. PMID 28453823